CLINICAL TRIAL: NCT00845676
Title: Treatment of Acute Hepatitis C Virus in HIV Co-Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California HIV/AIDS Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRP ID06-SF-218
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis C; Human Immunodeficiency Virus; HIV Infections
Keywords: Hepatitis C virus; Acute hepatitis C infection; HIV; HCV
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegylated interferon alfa-2a + Ribavirin (Experimental): Pegylated interferon alfa-2a + Ribavirin
  Interventions: Drug: Pegylated interferon alfa-2a + Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a + Ribavirin — Pegylated interferon alfa-2a 180 mcg subcutaneous injection once weekly for 24 weeks Ribavirin 1000-1200mg daily, dosed according to body weight and divided twice daily, for 12-24 weeks
  Other Names: Pegasys; PEG-IFN; RBV

SUMMARY:
This study is designed to test the hypothesis that treatment of hepatitis C virus (HCV) infection during the first 6 months after acquiring HCV among people who already have pre-existing HIV infection will result in improved responses to HCV therapy with a shorter duration of infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is one of the most important causes of illness and death among people living with HIV/AIDS. Over 200,000 people in the Unites States, including 37,000 in California, are co-infected with HIV and HCV. In the past, people who had both HIV and HCV often died from AIDS before HCV could cause serious problems. However, with improvements in HIV/AIDS care and treatment, more co-infected people are living longer and thus developing complications from their HCV, including liver scarring (called cirrhosis) and death. HCV infection can also make HIV medications more toxic to the liver, limiting HIV treatment options. Treatment for chronic (or long-term) HCV infection has improved in recent years, but people with HIV are still about half as likely to clear their chronic HCV infection with treatment as HIV-negative individuals. Also, HCV treatment can be very toxic and may have serious side effects for patients, particularly those with HIV.

Recent research suggests that treatment started within the first few months after getting HCV infection (called "acute infection") can result in high treatment response rates for people who do not have HIV. It is not known whether similarly high treatment response rates can also be seen in people with HIV. It has also been shown that each individual's response to the early phases of HCV treatment can predict his or her ability to clear HCV infection after the end of treatment. This study will look at whether it is possible to follow each person's own HCV viral load over time as a measure of treatment success and to tailor each individual's treatment to his or her own response. This idea is called "kinetically guided therapy" and is a new way of individualizing treatment regimen to produce high treatment success rates while minimizing the amount of potentially toxic medications that an individual might not need.

In this pilot study, 20 HIV-infected individuals with acute HCV infection will be treated with HCV therapy for 24 weeks. Because HIV co-infection decreases treatment success in chronic HCV infection, treatment will be started with the strong combination of pegylated-interferon plus ribavirin. However, this protocol will monitor each individual's HCV viral load during the first 12 weeks of treatment and will stop the ribavirin at week 12 if the individual has a good early response and might not need to continue both medications. Using this approach, pegylated interferon will be given for the full 24 weeks of treatment, but ribavirin will be continued for either 12 or 24 weeks, depending on each individual's early response to therapy. The primary endpoint for this study is the percentage of people who have a sustained virologic response to the study treatment. The side effects of treatment will also be measured in order to determine the overall risks and benefits of this approach to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly acquired HCV infection of 6 months or less duration
* Detectable HCV RNA at study entry
* HIV infection, any CD4 count

Exclusion Criteria:

* Pregnant or intent to become pregnant within 24 weeks of study completion
* Uncontrolled depression
* Other serious liver disease
* Other safety parameters must be met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hare, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital/UCSF, San Francisco, California, United States

REFERENCES:
- See also: Home page of the Positive Health Program, UCSF HIV/AIDS Division at San Francisco General Hospital — http://php.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at one U.S. clinical site
Groups:
- Experimental: Pegylated Interferon Alfa-2a + Ribavirin: Combination therapy with open-label pegylated interferon alfa-2a (PEG-IFN) + ribavirin (RBV): Pegylated interferon alfa-2a 180 mcg subcutaneous injection once weekly for 24 weeks. Ribavirin 1000-1200mg daily, dosed according to body weight and divided twice daily, for 12-24 weeks.
Period: Overall Study
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Started | 21
Completed | 19
Not Completed | 2
Not completed — Virologic breakthrough at week 20 | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 42 [26 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR)
Description: Proportion of subjects achieving a sustained virologic response (SVR), defined as undetectable HCV RNA 24-weeks after completion of treatment
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 19
percentage of participants | 62

2. Secondary Outcome: Safety and Tolerability of Treatment
Description: Number of participants with treatment-associated problems
Time Frame: 48 weeks
Population: PI left institution and sincere efforts were made to contact the PI, but were unsuccessful. No data are available to report.
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 0

3. Secondary Outcome: Association of SVR With Entry HCV RNA, Entry ALT, Entry CD4, and IL28B Genotype
Description: Predictors of SVR, including early HCV RNA response to treatment as they relate to SVR
Time Frame: 24 weeks
Population: as for outcome 2
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Experimental: Pegylated Interferon Alfa-2a + Ribavirin
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 13/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Pegylated Interferon Alfa-2a + Ribavirin (N=21)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
Virologic breakthrough (Infections and infestations) | 1 (1)
anemia (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes